CLINICAL TRIAL: NCT03093896
Title: The Effect of Consumption of Almonds and Snack Mix Daily for 6 Months on Performance on a Battery of Computerized Cognitive Tests (CANTAB) in Older Adults
Brief Title: The Effect of Consumption of Almonds and Snack Mix Daily for 6 Months on Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Elizabeth Johnson, Scientist I/Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 003
Record Dates: First submitted 2015-08-25; First posted 2017-03-28 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Mild Cognitive Impairment
Keywords: almonds; cereal snack
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- snack mix (Placebo Comparator): snack mix, 3 ounces: dried coconut, meat jerky, butter, cereal party mix
  Interventions: Dietary Supplement: snack mix
- almonds, 1.5 ounces (Active Comparator): almonds, 1.5 ounces/day
  Interventions: Dietary Supplement: almonds, 1.5 oz
- almonds, 3 ounces (Active Comparator): almonds, 3 ounces/day
  Interventions: Dietary Supplement: almonds, 3 oz

INTERVENTIONS:
Dietary Supplement: snack mix — commercial cereal mix with bits of beef jerky and coconut
  Arms: snack mix
Dietary Supplement: almonds, 1.5 oz — almonds, 1.5 oz/day
  Arms: almonds, 1.5 ounces
Dietary Supplement: almonds, 3 oz — almonds, 3.0 oz/day
  Other Names: almonds, 3.0 oz
  Arms: almonds, 3 ounces

SUMMARY:
Cognitive impairment is also a major risk factor for development of dementia later in life. Findings from recent studies suggest that the there are many nutrients contained in foods that may be important in cognitive function in the elderly. This study evaluates long-term intervention with almonds and snack mix as a treatment strategy for age-related cognitive impairment which could possibly prevent the onset of dementia.

The proposed study is designed as a randomized, placebo controlled trial that tests the effects of 6 month supplementation with 1.5 or 3 ounces of almonds or 3 ounces of shortbread containing coconut oil on cognitive function in older adults. Secondary outcomes include plasma biomarkers of oxidative stress and inflammation.

DETAILED DESCRIPTION:
The study is designed as a controlled trial that tests the effects of 6 month supplementation with 1.5 or 3 ounces of almonds or 3 ounces of snack mix a day on cognitive function in older adults. Subjects will be randomly assigned to one of the three groups. Secondary outcomes include plasma biomarkers of oxidative stress and inflammation. Participants will be recruited from community-dwelling men and women aged greater than of equal to 50 yr and less than or equal to 75 years and potential participants will be screened to meet cognitive and functional criteria. Participants will be pre-screened by telephone; those who appear to meet criteria will undergo further screening.

ELIGIBILITY:
Inclusion Criteria:

* men and women age >50 - 75 years
* body mass index >25-35 kg/m2
* Mini mental state exam (MMSE) score >24
* must be able to give written informed consent

Exclusion Criteria:

* history of active small bowel disease or resection
* atrophic gastritis
* uncontrolled blood pressure or untreated hypertension alcoholism (>2 drinks/d or 14 drinks/week)
* abnormal hematologic parameters that are determined by the study MD to influence study outcomes.
* endocrine disorders including diabetes or current pharmacological treatment of diabetes and untreated thyroid disease
* pancreatic disease
* anemia, and bleeding disorders
* nut allergy
* major chronic illness that might interfere with the study outcomes
* active cancer except for prostate cancer or cancer-free for at least 5 years
* unwilling to not use lutein, n3 fatty acid, or choline supplements for 2 months prior to study start
* diseases that interfere with fat absorption, e.g. colitis, celiac disease, Crohn's disease, cystic fibrosis (as determined by screening interview)
* rheumatologic diseases including gout or inflammatory arthritis
* immune deficiency conditions including autoimmune dieases, human immune deficiency virus (HIV); history of organ transplantation
* medications that interfere with fat absorption, e.g. bile sequestrants (as determined by screening interview)
* use of antipsychotic, antimanic, anti-inflammatory (except for aspirin and non steroidal anti-inflammatory drugs[NSAIDS]), monoamine inhibitors, or dementia medications
* inability to discontinue aspirin, NSAIDS for 72 hours prior to and for the duration of testing at study visits (baseline, 3 and 6 months)
* daily intake of proton pump inhibitors or H2 blockers
* smoking or use of nicotine patches or gum (within past 6 months)
* use of drugs suspected of interfering with metabolism of blood clotting with the exception of aspirin and NSAIDS, e.g. warfarin (as determined by screening interview)
* stroke, head injury with loss of consciousness or seizures.
* history or clinical manifestation of any significant neurologic disorder in the opinion of the investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2018-09 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
executive function executive function assessed by test administered via CANTAB (www.cambridgecognition.com) | change from baseline executive function at 6 months
  tests administered via CANTAB (www.cambridgecognition.com)

SECONDARY OUTCOMES:
attention assessed by test administered via CANTAB (www.cambridgecognition.com) | change from baseline attention at 6 months
  test administered via CANTAB (www.cambridgecognition.com)
visual memory assessed by test administered via CANTAB (www.cambridgecognition.com) | change from baseline visual memory at 6 months
  test administered via CANTAB (www.cambridgecognition.com)
inflammation - serum C-reactive protein as measured by ELISA kit | change from baseline serum CRP concentration at 6 months
  serum C-reactive protein - ELISA kit
inflammation - serum IL6 as measured by ELISA kit | change from baseline serum IL-6 concentration at 6 months
  serum IL-6 - ELISA kit
inflammation - serum IL12 as measured by ELISA kit | change from baseline serum IL-12 concentration at 6 months
  serum IL12 - ELISA kit
inflammation - serum ICAM as measured by ELISA kit | change from baseline serum ICAM concentration at 6 months
  serum ICAM - ELISA kit
plasma fatty acids | change from baseline plasma fatty acids concentration at 6 months
  measured by gas chromatography
plasma alpha-tocopherol | change from baseline plasma alpha-tocopherol concentration at 6 months
  measured by high pressure liquid chromatography
plasma magnesium | change from baseline plasma magnesium concentration at 6 months
  measured by atomic emission spectroscopy
fatty acids in red blood cells | change from baseline fatty acids concentration in red blood cells at 6 months
  measured by gas chromatography/mass spectroscopy
oxidative stress - aminothiols | change from baseline serum aminothiols at 6 months
  serum aminothiols - HPLC
oxidative stress - isoprostanes | change from baseline urinary isoprostanes at 6 months
  urinary isoprostanes - spectrophotometer
oxidative stress - superoxide dismutase | change from baseline serum superoxide dismutase at 6 months
  serum superoxide dismutase - ELISA kit
oxidative stress - glutathione peroxidase | change from baseline serum glutathione peroxidase at 6 months
  serum glutathione peroxidase - ELISA kit
oxidative stress - glutathione reductase | change from baseline serum glutathione reductase at 6 months
  serum glutathione reductase - ELISA kti
total serum cholesterol | change from baseline total serum cholesterol at 6 months
  colormetric assay Beckman Coulter AU400
serum low density lipoprotein | change from baseline serum low density lipoprotein at 6 months
  colormetric assay Beckman Coulter AU400
serum high density lipoprotein | change from baseline serum high density lipoprotein at 6 months
  colormetric assay Beckman Coulter AU400
serum very low density lipoprotein | change from baseline serum very low density lipoprotein at 6 months
  colormetric assay Beckman Coulter AU400

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Johnson, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mustra Rakic J, Tanprasertsuk J, Scott TM, Rasmussen HM, Mohn ES, Chen CO, Johnson EJ. Effects of daily almond consumption for six months on cognitive measures in healthy middle-aged to older adults: a randomized control trial. Nutr Neurosci. 2022 Jul;25(7):1466-1476. doi: 10.1080/1028415X.2020.1868805. Epub 2021 Jan 15. PMID 33448906